CLINICAL TRIAL: NCT04057716
Title: Eating-related Self-regulation and Its Neural Substrates as Mechanisms Underlying the Sleep/Eating Behavior Association in Children With Overweight/Obesity: An Ecological Momentary Assessment Study
Brief Title: Project REST: Regulation of Eating and Sleep Topography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andrea Goldschmidt, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY21070047; R01HL147914 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Childhood; Binge Eating; Sleep; Self-regulation
MeSH Terms: conditions — Pediatric Obesity; Bulimia; Self-Control

STUDY DESIGN:
Intervention Model Description: Participants will be instructed to restrict or expand their sleep for one week each within a randomized crossover design, separated by a one week wash-out period.
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to sleep condition in order to obtain unbiased estimates of study outcomes (e.g., weight, eating behavior).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep restriction followed by extension (Experimental): Children will spend 8 hours in bed for one week, engage in one week of wash-out, and then spend 11 hours in bed for one week.
  Interventions: Behavioral: Sleep restriction; Behavioral: Sleep extension
- Sleep extension followed by restriction (Experimental): Children will spend 11 hours in bed for one week, engage in one week of wash-out, and then spend 8 hours in bed for one week.
  Interventions: Behavioral: Sleep restriction; Behavioral: Sleep extension

INTERVENTIONS:
Behavioral: Sleep restriction — Participants will be asked to restrict their time in bed to 8 hours each night for one week.
  Other Names: Shortened sleep
Behavioral: Sleep extension — Participants will be asked to extend their time in bed to 11 hours each night for one week.
  Other Names: Extended sleep

SUMMARY:
Overweight/obesity and inadequate sleep are prevalent, and frequently co-occurring, health risks among children, both of which are associated with serious medical and psychosocial health complications including risk for cardiovascular disease. Although the investigator's data suggest that disrupted or shortened sleep may be causally associated with increased energy intake and weight gain in children, and with self-regulation and neural response to food cues in adults, understanding of mechanisms involved in the sleep/eating association is incomplete, thereby impeding development of targeted, optimally timed intervention strategies. The proposed mechanistic clinical trial aims to assess the effects of an experimental sleep manipulation on eating-related self-regulation and its neural substrates, and on real-world eating behavior, among children with overweight/obesity, which will help guide research efforts towards the refinement of prevention and intervention strategies targeting sleep and its eating-related correlates to curb weight gain throughout development.

DETAILED DESCRIPTION:
Insufficient sleep and excess weight status contribute to adverse health outcomes across the lifespan, including risk for cardiometabolic disease. Cross-sectional data suggest that children with overweight/obesity are more likely to experience sleep disturbances than their non-overweight peers. Although the nature of this association may be bidirectional, prospective studies indicate that sleep impacts body weight regulation through multiple physiological and psychological pathways. In particular, insufficient sleep is related to greater energy intake and reduced diet quality in children. Although mechanisms explaining the association between sleep and eating behavior are poorly understood, sleep restriction has been found to impact brain processes related to reward valuation of food and self-regulation, the behavioral manifestations of which may increase susceptibility to suboptimal dietary behaviors and subsequent weight gain. A limitation of prior research on mechanisms is that much of it has been conducted in adults and in laboratory settings, thereby calling into question the ecological validity of the findings. Alternatively, studies on sleep restriction/extension in children's natural environments have relied on retrospective reporting of eating behavior, included children across the weight spectrum, and had limited focus on underlying mechanisms, particularly neural substrates. A clearer understanding of momentary mechanisms involved in the sleep/eating association could improve development and/or refinement of sleep-related interventions, particularly those delivered in real time when risk for engaging in maladaptive eating is highest. The proposed R01 study will examine prospective associations among sleep, eating-related self-regulation, and eating behavior in the natural environment. Community-based children with overweight or obesity (n=120) will undergo a naturalistic protocol involving assessment of typical sleep and eating patterns (week 1), followed by sleep restriction or extension (weeks 2 and 3, separated by a 7-day wash-out), the latter occurring within a randomized crossover design. Assessment throughout the study period will involve daily actigraphy measurement of sleep patterns; repeated daily self-reports on eating behavior and behavioral assessment of eating-related self-regulation; and intermittent 24-hour dietary recalls informed by daily real-time food photography. Participants will complete fMRI-based assessment of neural activation during an eating-related self-regulation task after each week-long period of sleep restriction and extension. Overall aims are to assess short-term effects of sleep extension versus restriction on eating-related self-regulation (including behavioral and neural performance) and naturalistic eating behavior. These data will clarify timing and trajectory of changes in eating behavior and self-regulatory mechanisms as a consequence of sleep patterns. The proposed study has clear potential to advance scientific and clinical understanding of mechanisms involved in the prospective associations between inadequate sleep and maladaptive eating in youth and inform interventions to alleviate their cumulative personal and societal burden.

ELIGIBILITY:
Inclusion Criteria:

* at risk for obesity (BMI>=85th percentile for age and sex OR BMI>=50th percentile for age and sex with at least one obese parent)
* average time in bed between 9.5-10.5 hours/night

Exclusion Criteria:

* previous eating disorder diagnosis and/or sleep or psychiatric conditions
* conditions affecting executive functioning (e.g., recent concussion, traumatic brain injury)
* taking medication known to affect sleep/appetite (e.g., antihistamines, stimulants)
* receiving concurrent treatment for sleep or overweight/obesity

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Change in Weight Status | 4 weeks
  BMI (body mass index)
Change in Eating Behavior | 4 weeks
  measured by 24-hour dietary recall
Change in Eating Behavior | 4 weeks
  measured by ecological momentary assessment
Self-Regulatory Control | 4 weeks
  as measured by the Go/No-Go task (errors and response latency)

SECONDARY OUTCOMES:
Sleep Patterns | 2 weeks
  as measured by actigraph data

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Goldschmidt, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Weight Control & Diabetes Research Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lab website with description of current studies (including Project REST) — https://bite.pitt.edu/current-studies

DOCUMENTS (1):
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT04057716/ICF_003.pdf